CLINICAL TRIAL: NCT02229799
Title: Protocol for Post Marketing Surveillance of Actilyse Vial
Status: Terminated | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 135.315
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Stroke patients
  Interventions: Drug: Actilyse

INTERVENTIONS:
Drug: Actilyse

SUMMARY:
The objectives of this study are to review the safety and efficacy of Actilyse Vial (hereafter referred to as "Actilyse") in post-marketing use for treatment of acute ischemic stroke, through investigating followings;

1. Unknown adverse events (especially serious adverse events)
2. Frequency (Incidence) and trend of adverse events under the actual practice
3. Factors on the safety profile of Actilyse
4. Factors on the efficacy profile of Actilyse

ELIGIBILITY:
Inclusion Criteria:

* All in/out patients diagnosed as acute ischemic stroke

Exclusion Criteria:

1. Actilyse should not be administered to patients with high risk as follows:

   * Significant bleeding disorder at present or within the past 6 months, known hemorrhagic diathesis
   * Patients receiving oral anticoagulants, e.g. warfarin sodium (INR > 1.3)
   * Manifest bleeding or recent severe or dangerous bleeding
   * History or evidence or suspicion of intracranial hemorrhage including sub-arachnoid hemorrhage
   * Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
   * Hemorrhagic retinopathy (e.g. in diabetes, vision disturbances may indicate hemorrhagic retinopathy) or other hemorrhagic ophthalmic conditions
   * Prolonged or traumatic cardiopulmonary resuscitation (> 2 minutes), obstetrical delivery, within the past 10 days, recent puncture of a non-compressible blood-vessel (e.g. subclavian or jugular vein puncture)
   * Severe uncontrolled arterial hypertension
   * Bacterial endocarditis or pericarditis
   * Acute pancreatitis
   * Documented ulcerative gastrointestinal disease within the past 3 months, oesophageal varices, arterial-aneurysms, or arterial/venous malformations
   * Neoplasm with increased bleeding risk
   * Severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis
   * Hypersensitive to the active substance alteplase or to any of the excipients
2. In cases of acute myocardial infarction and acute pulmonary embolism, any history of stroke should be contraindicated.
3. In case that Actilyse is administered to acute ischaemic stroke, the followings should be contraindicated:

   * Symptoms of ischemic attack began more than 3 hours prior to infusion start or when time of symptom onset is unknown,
   * Symptoms of acute ischemic stroke that were either rapidly improving or only minor before start of infusion
   * Severe stroke as assessed clinically and/or by appropriate imaging techniques,
   * Seizure at onset of stroke
   * Evidence of intracranial hemorrhage (ICH) on the CT-scan
   * Symptoms suggestive of subarachnoid hemorrhage, even if CT-scan is normal
   * Administration of heparin within 48 hours preceding the onset of stroke with an elevated activated partial thromboplastin time (aPTT) at presentation
   * A combination of previous stroke and diabetes mellitus
   * Prior stroke or head trauma within the past 3 months
   * Platelet count of less than 100,000/mm3
   * Systolic blood pressure>185 mm Hg, or diastolic blood pressure>110 mm Hg, or aggressive management (IV medication) is necessary to reduce blood pressure to these limits
   * Blood glucose<50mg/dl or >400 mg/dl
4. Acute stroke patients between the age of ≤ 18 or ≥ 80 years

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2003-02; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness assessed by 30 days-mortality | 30 days
Number of patients with adverse events | up to 30 days
Number of patients with clinically significant abnormal findings in physical examination | up to 30 days